CLINICAL TRIAL: NCT04039906
Title: A Single-institutional Study to Assess the Impact of ANDY(Automatic Needle Destroyer) to the Medical Staffs in Terms of Working Efficiency Assessed by Working Time and Satisfaction Assessed by Usability and Safety Using SUS Score and Survey
Brief Title: A Single-institutional Study to Assess the Time Efficiency and Working Satisfaction Using ANDY(Automatic Needle Destroyer)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-05-112
Record Dates: First submitted 2019-07-15; First posted 2019-07-31 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-05

CONDITIONS: Needle Stick Injuries
Keywords: Efficiency,Usability,Safety
MeSH Terms: conditions — Needlestick Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Removal of needle with existing method (No Intervention): Participants will remove needles from syringes with the existing method like they are already doing. (Record the time required for the needle removal procedure by photographing during 24 hours/7 days.)
- Removal of needle with using ANDYs (Experimental): Participants will remove needles from syringes with Andy. (Record the time required for the needle removal procedure by photographing during 24 hours/7 days.)
  Interventions: Device: Removal of needle with using ANDYs

INTERVENTIONS:
Device: Removal of needle with using ANDYs — 1. ANDY will be provided to medical staffs to be use in removal needles from syringes during 7 days
  2. Record the time required for the needle removal procedure by photographing the needle removal procedure during 24 hours/7 days.
     Identify the number of syringes processed by ANDY.
  3. After 3rd week, do survey and interview 15 people selected by the convenient sample method. By interviewing, collect information of overall experience after using automated needle processing system, how long their hospital working experience is, and other information or systems the interviewees felt those are necessary.
  Arms: Removal of needle with using ANDYs

SUMMARY:
Evaluate the efficiency of adopting the automated needle processing system by evaluating efficiency, usability and safety when using ANDY(Automatic Needle Destroyer). Install ANDY(Automatic Needle Destroyer) in the ER, and evaluate the system by comparing the efficiency of the work, usability, actual decrease ratio of needlestick injury between using the automated needle processing system and not using it.

DETAILED DESCRIPTION:
1. Background The most frequent occupational injury is exposure to blood and fluid by needlestick injury. Needlestick injuries can result in serious infections if appropriate infection control measures are not taken promptly.

   Since the use of safety devices are not popularly used, the needle and syringe are mostly taken into pieces by physical ways. There are some cases that the needle and syringe is not separated, and the entire syringe can be put directly into the waste container. There is also a problem that it takes a lot of time and efforts to remove needles from syringes. In addition, the existing safety mechanism is physical methods such as pulling out the needle, damaging or cutting the needle, or using heat to the needle, or melting it by using chemicals. It is a semi-manual since you have to wait holding the syringe during the process, and it is inconvenient to use considering a busy medical environment.

   Therefore, we developed ANDY(Automatic Needle Destroyer) that can be introduced at a convenient and reasonable cost, and try to objectively evaluate the utility of ANDY in a clinical environment.
2. Purpose The purpose of this study is to Evaluate the efficiency of adopting the automated needle processing system by evaluating efficiency, usability and safety of the system.
3. Design : RCT (randomized controlled trial)
4. Setting: EMERGENCY CENTER at the Samsung Medical Center
5. Enrollment : 129 medical staffs in the ER. 10ea ANDY and 10ea of Existing waste containers(needle box)
6. Intervention :

   6-1) 1st Week : Removal of needle with existing method
   * Record the time required for the needle removal procedure by photographing the needle removal procedure during 24 hours/7 days.
   * Identify the number of syringes processed by existing method.
   * Do survey after 1st week

   6-2) 2nd week: Prepare for using ANDYs
   * Provide clinicians with instruction how to use ANDY
   * Install 10 ANDYs in the ER.

   6-3) 3rd week : Removal of needle with using ANDYs
   * Record the time required for the needle removal procedure by photographing the needle removal procedure during 24 hours/7 days.
   * Identify the number of syringes processed by ANDY.
   * After 3rd week, do survey and interview 15 people selected by the convenient sample method. By interviewing, collect information of overall experience after using automated needle processing system, how long their hospital working experience is, and other information or systems the interviewees feel those are necessary.
7. Scoring: By the answers of the Questionnaire of Satisfaction (SUS and adjective score)
8. Study period : 3 weeks
9. Satisfaction survey: SUS and adjective score

ELIGIBILITY:
Inclusion Criteria:

* medical staff of the ER
* adult ER medical staff over 19 years of age
* A subject who voluntarily agrees and signs

Exclusion Criteria:

•A subject who did not agree with this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Time Efficiency: Comparing the time required to remove the needle from syringe for assessing change in time between using automated needle processing system or not | [1st Week] : Removal of needle in accordance with existing method, [3rd week] : using a ANDY(automated needle processing system)
  - Comparison of the required time(second) to remove the needle between using the automated needle processing system and not using it.

SECONDARY OUTCOMES:
Usability: Comparing the SUS score for assessing the change in usability between using automated needle processing system or not | [1st Week] : Removal of needle in accordance with existing method, [3rd week] : using a ANDY(automated needle processing system)
  - Comparison of the usability between using the automated needle processing system and not using it by doing survey after 1st week and 3rd week and Interview after 3rd week( Scoring by the answers of the Questionnaire of Satisfaction (SUS) and adjective score)
Safety: Comparing the number of accidents of the needlestick injuries between using automated needle processing system or not | [1st Week] : Removal of needle in accordance with existing method, [3rd week] : using a ANDY(automated needle processing system)
  - Comparison of the number of accidents of the needlestick injuries between using the automated needle processing system and not using it.

CONTACTS AND LOCATIONS:
Overall Officials: TAERIM KIM, Doctoral, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided